CLINICAL TRIAL: NCT02682290
Title: Assessment of a Device Used for Measuring the Rheological Parameters of Human Sputum.
Brief Title: Assessment of Rheological Parameters of Human Sputum.
Acronym: RHEOMUCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 38RC14.444
Record Dates: First submitted 2016-01-27; First posted 2016-02-15 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: COPD; Asthma; Cystic Fibrosis
Keywords: SPUTUM; RHEOLOGY
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rheological measurement of sputum (Other): patients with COPD and patient with cystic fibrosis will perform a spontaneous expectoration.
  Then all participants will have an induced expectoration with hypertonic salin solution.
  Interventions: Other: Expectoration and measurement of sputum rheological properties

INTERVENTIONS:
Other: Expectoration and measurement of sputum rheological properties

SUMMARY:
This is a proof of concept study. The aim of this study is to assess a device measuring rheological properties of human sputum of four populations :

* 10 patients with Broncho Chronic Obstructive Pulmonary Disease (COPD)
* 10 patients with asthma
* 10 patients with cystic fibrosis
* 10 healthy volunteers.

DETAILED DESCRIPTION:
This study includes two visits to 48 hours apart.

During the first visit :

* Patients with COPD or cystic fibrosis will have a spontaneous expectoration
* Then all study participants will have an induced expectoration with hypertonic salin solution (4.5%).

During the second visit :

* Patients with COPD or cystic fibrosis will have a spontaneous expectoration
* Then, patients with COPD, asthma and healthy volunteers will have an induced expectoration with hypertonic salin solution (4.5%). Patients with cystic fibrosis will have a spontaneous expectoration 1 hour after an RhDNAse nebulization.

A control spirometry will be perform before each expectoration and during induced expectoration if necessary.

All sputum sample collected will be homogenized and then divided into two equal volumes in order to perform two separate rheological measurements of 15 minutes.

ELIGIBILITY:
Inclusion Criteria of healthy volunteers:

* 18>BMI>29
* No smoker
* No acute disease in the previous month

Exclusion Criteria of healthy volunteers:

* asthma, COPD, cystic fibrosis
* contraindications for spirometry
* pregnant woman
* legal exclusion criteria

Inclusion Criteria of patients with cystic fibrosis:

- cystic fibrosis with bronchial disorder. Diagnosis confirmed by a reference center

Exclusion Criteria of patients with cystic fibrosis:

* Forced Expiratory Volume in 1 second (FEV1 ) ≤ 40%, contraindications for RhDNAse, patient with chronic impairment of lung function (PaO2<60 mmHg at rest). Patient who is unable to perform a spontaneous expectoration.
* case of acute exacerbation during the last month
* contraindications for spirometry
* pregnant woman
* legal exclusion criteria

Inclusion Criteria of patients with COPD:

- COPD with FEV1/Forced Vital Capacity (FVC) <70% after administration of a beta-2 agonist

Exclusion Criteria of patients with COPD:

* Patient with chronic impairment of lung function and/or FEV1≤ 40%. Patient who is unable to perform a spontaneous expectoration.
* case of acute exacerbation during the last month
* contraindications for spirometry
* pregnant woman
* legal exclusion criteria

Inclusion Criteria of patients with asthma:

- diagnosis of asthma confirmed by a Pulmonologist

Exclusion Criteria of patients with COPD:

* Patient with chronic impairment of lung function and/or FEV1≤ 50%.
* Very unstable Asthma
* case of acute exacerbation during the last month
* contraindications for spirometry
* pregnant woman
* legal exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2017-07-04 (Actual)

PRIMARY OUTCOMES:
Reproducibility of the rheological measurements of human sputum | Day1 (at the first visit)
  The reproducibility will be assessed during the first visit (Day1). The two rheological measurements performed 15 minutes apart will be compared.
  Rheological measurements : elastic modulus G' at 0.7Hz, elastic modulus G' at 3Hz, viscous modulus G'' at 0.7Hz, viscous modulus G'' at 3Hz)

SECONDARY OUTCOMES:
Reproducibility of the rheological measurements of human sputum | Day3 (48h00 after day1)
  Comparison between the average of the two rheological measurements preformed at the first visit (Day1) and the average of the two rheological measurements preformed at the second visit (day3) 48 hours later.
Feasibility of the rheological measurements | Day1 (at the first visit) and day3 (48h00 after day1)
  frequency of measurements failure
Comparison of sputum rheological measurements between the four populations studied (healthy volunteers, Asthma, COPD, Cystic Fibrosis) | Day1 (at the first visit) and day3 (48h00 after day1)
Influence of two mucolytic treatments (hypertonic saline solution, RhDNAse) on rheological measurements of patient with cystic fibrosis | Day1 (at the first visit) and day3 (48h00 after day1)
  During the first visit (day1), for patients with cystic fibrosis: Comparison of rheological parameters before and after nebulization of saline solution.
  During second visit (day 3) for patients with cystic fibrosis: Comparison of rheological parameters before and after nebulization of 2.5 ml of RhDNAse.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Investigation Clinique - INSERM 1406, Grenoble, Isere, France

IPD SHARING:
Plan to Share IPD: No